CLINICAL TRIAL: NCT00260728
Title: ACCESS: Prospective, Multi-center Trial of the Fusion Vascular Access Graft for Patients Who Require Early Vascular Access for Hemodialysis
Brief Title: The Boston Scientific ACCESS Trial
Acronym: ACCESS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Maquet Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2100; G050151
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Renal Disease; Kidney Failure
Keywords: vascular access; hemodialysis
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Device: vascular access graft implantation

INTERVENTIONS:
Device: vascular access graft implantation — vascular access graft implantation

SUMMARY:
The Boston Scientific ACCESS trial seeks to study the safety and to evaluate the success of the Fusion™ Vascular Access Graft for patients in need of early vascular access for hemodialysis.

DETAILED DESCRIPTION:
The Boston Scientific ACCESS trial seeks to study the safety and to evaluate the success of the Fusion™ Vascular Access Graft for patients in need of early vascular access for hemodialysis. The primary objective is to demonstrate that secondary patency at 6 months for the Fusion™ Vascular Access Graft is not less than an objective performance criterion (OPC) minus a clinically relevant margin (δ). The OPC represents secondary patency at 6 months for the standard of care access grafts.

The secondary safety endpoint is the occurrence of CEC-adjudicated device or procedure related adverse events through 24 months post implant procedure, or through discharge for patients with unsuccessful device implantation. Secondary efficacy endpoints include:primary patency; primary assisted patency; ability to revise a failed graft; early access capability; time to hemostasis.

Subjects will undergo a thorough medical assessment and physical examination pre-procedure and will be assessed peri-procedure. Enrolled subjects with a device implanted will be evaluated at 1, 6, 12, 18 and 24 months post implant procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Need for early dialysis access (≤72 hours after implantation):

   * Initiation of maintenance dialysis is recommended per K/DOQI or institutional guidelines; or
   * Patient is currently receiving dialysis via catheter
2. No prior implantation of synthetic graft in the arm to be treated
3. Life expectancy of at least 2 years, based on physician's assessment of medical condition

Exclusion Criteria:

1. Patient younger than 18 years of age
2. Any stenosis in the veins proximal to (downstream of) implant site, as determined previously or by current ultrasound
3. Pregnancy
4. Bleeding disorder, e.g., low platelet count (<50,000), hypercoagulable state, e.g., antithrombin III deficiency; antiphospholipid or anticardiolipin antibodies; Factor V Leiden; circulating Lupus anticoagulant; current, active heparin-induced thrombocytopenia; Protein C or S deficiency; or history of recurrent deep vein thrombosis not related to AV access.
5. Active malignancy, e.g., condition either being treated or considered untreatable
6. Active systemic infection, e.g., condition either being treated or considered untreatable
7. Uncontrolled major symptomatic medical problem, e.g., undiagnosed severe pain, metabolic disturbance, fever, etc.
8. Likelihood of poor compliance to required dialysis protocol, e.g., history of poor attendance to required clinic sessions or non-compliance to medication
9. Mental incapacity; inability to understand treatment instructions
10. Currently participating in another investigational drug or device study that clinically interferes with the endpoints of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2005-12; Primary Completion 2007-05 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Secondary patency at 6 months as determined by ability of the graft to be used for vascular access for hemodialysis | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Luis Sanchez, MD, Principal Investigator — Washington University School of Medicine, Barnes Jewish Hospital
Locations (8):
- United States (8):
  - Long Beach VA Medical Center, Long Beach, California
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - VA New Jersey Healthcare System, East Orange, New Jersey
  - New York - Presbyterian, Columbia University Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Texas Southwestern / VA Medical Center, Dallas, Texas